CLINICAL TRIAL: NCT07256730
Title: Comparative Study Between Artificial Intelligence-Assisted/Computer-Guided Versus Conventional Ridge Splitting Utilizing Electromagnetic Mallet for Reconstruction of Horizontal Ridge Defects: A Randomized Controlled Clinical Study
Brief Title: Computer-Guided Ridge Split and Expansion Using an Electromagnetic Mallet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Assistant Professor, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-338
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Reconstruction of Horizontal Ridge Defects
Keywords: ridge defects; ridge split; electromagnetic mallet; dental implant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freehand spit (Experimental): conventional ridge splitting with conventional simultaneous implant placement
  Interventions: Procedure: free-hand ridge splitting
- computer-guided split (Experimental): computer-guided ridge splitting assisted by artificial intelligence with simultaneous computer-guided implant placement.
  Interventions: Procedure: AI/guided ridge splitting

INTERVENTIONS:
Procedure: free-hand ridge splitting — Midcrestal incision will be followed by reflection of a full-thickness flap. A midcrestal cut without vertical osteotomy will be done using electromagnetic mallet unit, and then the cut will be extended deep to the implant length. The ridge will be expanded progressively using bone wedges. Dental implant fixtures will be placed stably with 1 mm minimal thickness of buccal bone plate. Surgical site will be completely closed, and wound edges will be sutured in a tension-free way.
  Arms: Freehand spit
Procedure: AI/guided ridge splitting — The patient specific guides will be placed and fixed by monocortical osteosynthesis screws at the pre-planned positions at the labial buccal mucosa.
  A midcrestal cut will be performed on the crest of the alveolar ridge guided by the guide slits. The cuts will be expanded progressively using bone wedges through the guide slits to gradually lateralize and expand the labial alveolar plate of bone, so the labial cortex will move through the intentionally created micro gap till it touches the fitting aspect of the patient-specific guide. Implant drills will be inserted through the guiding holes in the surgical guide, and the implant osteotomy sites will be prepared. Finally, implants will be inserted in the osteotomy sites using a torque wrench in a self-tapping fashion, engaging palatal and basal bone for primary stability.
  Arms: computer-guided split

SUMMARY:
The current trial aims to assess the efficacy of utilizing the electromagnetic mallet either by AI-assisted digital workflow or by the conventional freehand approach for reconstruction of horizontal ridge defects utilizing the ridge-split and expansion technique.

DETAILED DESCRIPTION:
Dental implants are a durable and long-term choice for tooth replacement to provide both functional and aesthetic benefits. However, successful implantation is critical, as it needs a sufficient amount of bone to maintain an ideal implant pathway and avoid vital structures. Vertical and horizontal ridge defects might occur after tooth extraction.

The pattern of alveolar ridge defect after extraction is classified according to the Cologne Classification into horizontal, vertical, combination, and sinus defects. mild (up to 4 mm), moderate (4-8 mm), and significant (over 8 mm) atrophy.

Successful implant placement is difficult to maintain with insufficient bone height and width. Many surgical techniques were introduced for the horizontally collapsed ridges, such as ridge augmentation, block graft, guided bone regeneration, and onlay graft. But these techniques need a long period of time for reconstruction, and an additional surgery is required for delayed implant placement.

Among these techniques, the ridge-splitting technique was performed for treating horizontally collapsed ridges by means of splitting the deficient ridge followed by ridge expansion to accommodate simultaneous implant placement.

The concept of the ridge-splitting technique is to make a self-space-making defect. The ridge-splitting technique was introduced by Tatum Jr. in 1986 and reintroduced in 1990 by Scipioni et al. In 1994, the technique was adapted by Summers, who utilized the viscoelastic properties of bone by applying pressure in-between buccal and lingual cortical bones using Summers osteotome to increase the width of the bone.

The ridge-splitting technique allowed the clinician to achieve desirable results within the shortest period and provide ridge expansion with simultaneous implant placement without the need for additional surgery and increase wound healing and satisfaction of the patient. Different instruments were used for splitting, such as chisels, discs, saws, osteomes, piezo surgery, and electromagnetic mallets.

The electromagnetic mallet consists of a handpiece that produces electromagnetic pulses with a rapid, non-impact motion that transmits to its tip, allowing high-intensity and precise movements with reduced trauma, minimal tissue damage, a greater safety margin, improved surgical outcomes, and faster recovery times. The precise movements make the repeatability of the procedure more applicable, which is very difficult to obtain with manual instruments.

Computer-guided surgery provides predictable and accurate treatment planning and implant positioning. It permits visualizing the jawbones and vital anatomical structures for preserving them during guided surgery. Artificial intelligence (AI) refers to the ability of machines to execute tasks that traditionally require human intelligence. Enhancing the high-quality dental treatment and precision of patient management, diagnosis, and treatment planning.

The current trial aims to assess the efficacy of utilizing the electromagnetic mallet either by AI-assisted digital workflow or by the conventional freehand approach for reconstruction of horizontal ridge defects utilizing the ridge-split and expansion technique.

ELIGIBILITY:
Inclusion Criteria:

1. The target population with inadequate bone volume for implant placement due to width insufficiency of maxillary anterior alveolar ridges.
2. Age ranges from 18 to 40 years of both sexes.
3. Absence of any complicating systemic condition that may contraindicate surgical procedures and implant placement.
4. Adequate oral hygiene.
5. Eligible participants should present good general health and agree to random assignment to any of the two parallel study groups.
6. Participants had a minimum 3-month post-extraction healing period and a horizontal defect in the maxillary esthetic zone with at least a bone width of 3 mm.

Exclusion Criteria:

1. Vertical ridge defect.
2. Undercut on the labial/buccal side.
3. Thick cortical bone without cancellous bone inside.
4. Uncontrolled systematic disorders as, diabetes mellitus, uncontrolled periodontal disease, history of head and neck radiotherapy, smokers, pregnancy, noncompliant patients, allergy to the used medications, uncooperative individuals or those unable to attend the study follow-up appointments.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
alveolar ridge width | 12 months
  CBCT will have taken immediately after surgery and at 6 and 12 months postoperatively

SECONDARY OUTCOMES:
vertical bone height | 12 months
  CBCT will be taken immediately after surgery and at 6 and 12 months postoperatively to evaluate vertical bone height.

CONTACTS AND LOCATIONS:
Overall Officials: walid elamrousy, Study Chair — Kafrelsheikh University
Locations (1):
- Faculty of Dentistry, Periodontology Department, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elayah SA, Younis H, Cui H, Liang X, Sakran KA, Alkadasi B, Al-Moraissi EA, Albadani M, Al-Okad W, Tu J, Na S. Alveolar ridge preservation in post-extraction sockets using concentrated growth factors: a split-mouth, randomized, controlled clinical trial. Front Endocrinol (Lausanne). 2023 May 17;14:1163696. doi: 10.3389/fendo.2023.1163696. eCollection 2023. PMID 37265705